CLINICAL TRIAL: NCT06446427
Title: The Effect of Acute High Altitude Exposure on Rescuer Performance and Patient Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024-00237
Record Dates: First submitted 2024-05-15; First posted 2024-06-06 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: High Altitude; Hypobaric Hypoxia; Risk Reduction
Keywords: High Altitude; Hypobaric Hypoxia; Patient Care; Patient Safety; Rescuer Safety; Emergency Medicine; Anaesthesia
MeSH Terms: conditions — Altitude Sickness; Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: The investigators imply a repeated measures design. A group of 20 participants will perform in simulated medical scenarios sequentially under four different circumstances (baseline, interventions 1-3)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants cannot be masked to whether they are at high or low altitude and whether they have spent a night at high altitude. However, they will not know whether they receive air (baseline, interventions 1 and 3) or supplementary oxygen nasally at the same flow rate (intervention 2).
  Outcome Assessors will be fully blinded. They assess the medical performance on video recordings of the simulated scenarios, and will not know which time point a specific scenario has taken place (baseline, interventions 1-3) and whether participants receive air or supplementary oxygen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Acute high altitude exposure — Thirty minutes after arrival at the Research Station Jungfraujoch by train, a simulated scenario of patient care ("intervention 1", high altitude at 3450 masl) is performed.
  Other Names: Intervention 1
Other: Acute high altitude exposure, with supplementary oxygen — 4 hours after arrival at the Research Station Jungfraujoch by train, a simulated scenario of patient care ("intervention 2", high altitude at 3450 masl) is performed, while the participants receive 4 litres / minute of oxygen via nasal route.
  Other Names: Intervention 2
Other: Subacute high altitude exposure, after having spent a night at high altitude — After having spent a night at the Research Station Jungfraujoch, a simulated scenario of patient care ("Intervention 3", high altitude at 3450 masl) is performed.
  Other Names: Intervention 3

SUMMARY:
Rescue services in mountainous regions are frequently called to missions at altitudes >3000 m. Under the difficult conditions of acute exposure to altitude, the crews then have to undertake demanding medical and rescue measures. Previous studies in non-medical personnel, such as astronauts, aircraft pilots, and military helicopter pilots have found that the lack of oxygen associated with acute exposure to altitude may impair cognitive functions. No data exists on the effect this may have on the performance of medical staff in terms of patient examination, communication, decision-making, planning, and overall patient care. This study aims to close this knowledge gap. The investigators of this study aim to make rescue missions to high altitude safer for both the patients and the rescuers.

To assess the effect of high altitude on patient care, the investigators recruit highly trained medical specialists who will perform patient care in simulated scenarios both at high altitude and at low altitude. These scenarios will be recorded and the performance of the medical specialists judged by independent reviewers.

The medical specialists will also perform in simulated scenarios at high altitude two more times: once with supplementary oxygen, and once after spending a night at high altitude. the investigators do this to evaluate whether supplementary oxygen improves their performance, and whether symptoms of acute mountain sickness (which usually develop after spending the first night at high altitude) decreases their performance further.

DETAILED DESCRIPTION:
Rescue services in mountainous regions are frequently called to missions at altitudes >3000 m. Under the difficult conditions of acute exposure to altitude, the crews then have to undertake demanding medical and rescue measures, such as an emergency induction of anaesthesia, resuscitation, treatment of polytraumatized patients, or a winch manoeuvre by helicopter in exposed, fall-prone terrain.

The exponential decrease in barometric pressure at altitude results in hypobaric hypoxia (HH), leading to a reduction in the partial pressure of oxygen at every point along the oxygen transport chain from the ambient air to tissue mitochondria. If the body's adaptive mechanisms fail to compensate for the lack of oxygen, symptoms like headache, nausea, fatigue, and dizziness may occur. In addition, HH may impair higher cortical functions. Individuals affected by high altitude frequently do not recognise a decline in cognitive function and overall performance, which can lead to incidents and even fatal consequences.

Previous studies in non-medical personnel, such as astronauts, aircraft pilots, and military helicopter pilots have explored the influence of HH on multiple cognitive domains. Impairment of working memory was described during hypoxia awareness trainings and in pilots while others reported no effects. Some studies have reported reduced psychomotor vigilance, while others found no effects. To counteract these impairments, the European Union Aviation Safety Agency (EASA) mandates simulated hypoxia training for pilots flying rescue missions to above 4000 m.

Studies in medical personnel are few and mostly focused on the quality of cardiopulmonary resuscitation (CPR) at (simulated) high altitude. High-quality CPR, which can be physically demanding for rescuers even under normoxic conditions, leads to rescuer fatigue faster under HH. Two recent studies have shown that HH leads to a lower quality of CPR at simulated and natural high altitude. A smaller study found simulated altitude to have a negative effect on the quality of ventilation but not on chest compression. A recent study reported a slower reaction time in medical personnel at simulated high altitude. Particularly noteworthy is the fact that rescuers did neither notice the reduced cognitive function nor the decreased quality of CPR they provided under HH, even though they were highly trained helicopter emergency medical services personnel. To the investigators' knowledge, CPR at high altitude has only been studied as an isolated skill. No data exist on the performance of medical staff in terms of patient examination, communication, decision-making, planning, and overall patient care. This study aims to close this knowledge gap. The findings of this study may help to broaden the understanding of HH, and lay the ground for further research in high altitude rescue.

As the primary endpoint of this study, the investigators evaluate medical performance and patient care using validated scores for medical skills and non-technical skills (Modified Simulation Team Assessment Tool (STAT), Concise Assessment of Leader Management (CALM), Team Emergency Assessment Measure (TEAM). These three scores are averaged (25% STAT, 25% CALM, 50% TEAM) to form a composite score. Scores are assessed by an analysis of video recordings of the simulated scenarios by independent outside assessors.

Secondary endpoints are described in detail elsewhere. They involve the measurement of reaction speed, risk assessment ability, cognitive function, the presence/absence of acute mountain sickness (AMS), the self-assessment of cognitive capacity, and basic vital functions. The concrete tests and measurements the investigators imply are:

* Psychomotor Vigilance Test (PVT)
* Balloon Analogue Risk Task (BART)
* Digit Symbol Substitution Test (DSST)
* Lake Louis Score (LLS), AMS is present at a score of three or higher
* Self-Assessment of Cognitive Capacity on a scale of 1-10
* Heart rate, Blood-pressure, peripheral blood oxygen saturation (SpO2) as measured by non-invasive means

The investigators will assess medical performance (and all other tests and measurements mentioned above) at four time points (baseline, interventions 1-3).

Testing at 30 minutes after arrival by train at high altitude (the High Altitude Research Station Jungfraujoch, 3450 m, "intervention 1") and at low altitude (Bern, 540 m, "baseline") are performed to answer the main hypothesis; whether acute rescuer exposure to high altitude impairs patient care.

To answer the additional research questions, additional testing will be performed at high altitude 4 hours after arrival with supplemental oxygen (4 litres/min, nasal) ("intervention 2") and after spending the night at 3450 m ("intervention 4").

At the four time points of measurement, the participants will have to run through one of the following four scenarios of simulated patient care:

1. A polytraumatised 35 y.o. patient who fell 12 metres. Adequate treatment will entail: anamnesis, immobilisation of the cervical spine, treatment of a tension pneumothorax, installation of analgosedation.
2. A 64 y.o. patient with acute abdominal pain and nausea due to an acute myocardial infarction. Adequate treatment will entail: Anamnesis, performing and interpreting a 12-lead electrocardiogram, resuscitation.
3. A 35 y.o. mother with her 5 m.o. child who is experiencing a seizure. Adequate treatment will entail: Anamnesis, treatment of the epileptic seizure, recognition of impeding respiratory failure and consequent assisted ventilation.
4. A 19 y.o. hypothermic patient. Adequate treatment will entail: Anamnesis, recognition of likely hypothermia and taking measures to avoid afterdrop, resuscitation according to hypothermia protocols, adequate care after return of spontaneous circulation.

All four scenarios are designed to be of equal difficulty. However, the order of the scenarios is randomised electronically before the start of the study, so that different participants go through different scenarios at all points of measurements (baseline, interventions 1-3). This is done to avoid skewing of performance due to some scenarios being inadvertently more difficult or easier than others.

Before each scenario, the participants undergo all tests and measurements outlined above (PVT, BART, DSST, LLS, Self-Assessment of Cognitive Capacity on a scale of 1-10, Heart rate, Blood-pressure, peripheral blood oxygen saturation).

Supplemental application of oxygen during intervention 2 might bias the participants. Therefore, they will receive air via nasal cannula at the same flow rate during all other scenarios (baseline, interventions 1 and 3) in the sense of a "placebo administration".

ELIGIBILITY:
Inclusion Criteria:

Medical doctors with certification and experience in preclinical emergency medicine, defined as (all must apply):

* 2 or more years of training in anaesthesiology
* 3 or more months of preclinical work
* 50 or more cases as the lead preclinical physician with potential danger to the patient's life (with a National Advisory Committee for Aeronautics score (NACA) of 4 or more)
* A valid preclinical certification (Swiss "Notarztkurs" or similar)
* Written informed consent to participate in the study

Exclusion Criteria (none must apply):

* Any medical condition known to place the participant at higher risk for hypoxia-induced adverse events (cardiovascular, pulmonary, neurological, otherwise).
* Pre-acclimatisation to high altitude, defined as travel to above 2500 m in the 4 weeks previous to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The effect of acute high altitude exposure on medical performance, measured by the STAT score | Baseline, intervention 1 (30 minutes after arriving at high altitude)
  The investigators asses the quality of patient care at low and high altitude exposure.
  The primary outcome of the study - a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT) - will be analysed by means of a linear mixed-effect regression model to account for the longitudinal study design. In particular, each of the four time points represents a fixed effect (implemented with a factor variable) and a random offset for each participants is included in the model allowing to represent the repeated measurements and associated covariance structure.
  The analysis of the primary endpoint - the difference in the composite score between baseline and after acute altitude exposure (intervention 1) - will be performed by assessing the pairwise contrast of the estimated marginal means of the linear mixed-effect regression model.
The effect of acute high altitude exposure on medical performance, measured by the CALM score | Baseline, intervention 1 (30 minutes after arriving at high altitude)
  The investigators asses the quality of patient care at low and high altitude exposure.
  The primary outcome of the study - a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT) - will be analysed by means of a linear mixed-effect regression model to account for the longitudinal study design. In particular, each of the four time points represents a fixed effect (implemented with a factor variable) and a random offset for each participants is included in the model allowing to represent the repeated measurements and associated covariance structure.
  The analysis of the primary endpoint - the difference in the composite score between baseline and after acute altitude exposure (intervention 1) - will be performed by assessing the pairwise contrast of the estimated marginal means of the linear mixed-effect regression model.
The effect of acute high altitude exposure on medical performance, measured by the TEAM score | Baseline, intervention 1 (30 minutes after arriving at high altitude)
  The investigators asses the quality of patient care at low and high altitude exposure.
  The primary outcome of the study - a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT) - will be analysed by means of a linear mixed-effect regression model to account for the longitudinal study design. In particular, each of the four time points represents a fixed effect (implemented with a factor variable) and a random offset for each participants is included in the model allowing to represent the repeated measurements and associated covariance structure.
  The analysis of the primary endpoint - the difference in the composite score between baseline and after acute altitude exposure (intervention 1) - will be performed by assessing the pairwise contrast of the estimated marginal means of the linear mixed-effect regression model.

SECONDARY OUTCOMES:
The effect of supplementary oxygen on medical performance during acute high altitude exposure, measured as a composite of STAT, CALM, and TEAM scores | Baseline, intervention 1 (30 minutes after arriving at high altitude), intervention 2 (4 hours after arriving at high altitude, with supplementary oxygen)
  The investigators asses any changes to the quality of patient care when participants receive supplementary oxygen during acute high altitude exposure. Since acute effects of high altitude exposure are mainly due to hypobaric hypoxia, supplementary oxygen might improve patient care. Patient care is measured through a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT).
  The investigators use the same linear mixed-effect regression model as described under the primary outcome for the assessment of this outcome, but comparing intervention 2 (4 hours after arrival at high altitude, with supplementary oxygen) to baseline) and intervention 1 (at 30 minutes after arrival at high altitude).
The effect of subacute high altitude exposure on medical performance, measured as a composite of STAT, CALM, and TEAM scores | Baseline, intervention 1 (30 minutes after arriving at high altitude), intervention 3 (after having spent a night at high altitude)
  The investigators asses the quality of patient care under subacute high altitude exposure, i.e. after having spent a night at high altitude. At the altitude at which the study takes place, 30-40% of participants are expected to develop mild to moderate symptoms of acute mountain sickness, which might impair the quality of patient care they provide. The presence and severity of AMS will be assessed by the Lake Louis Score. AMS is present at a score of 3 or higher. Patient care is measured through a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT).
  The investigators use the same linear mixed-effect regression model as described under the primary outcome for the assessment of this outcome, but comparing intervention 3 (after having spent a night at high altitude, no supplementary oxygen) to baseline and intervention 1 (at 30 minutes after arrival at high altitude).
The effect of gender and age on medical performance during low altitude, acute and subacute high altitude exposure, measured as a composite of STAT, CALM, and TEAM scores | Baseline, intervention 1 (30 minutes after arriving at high altitude), intervention 2 (4 hours after arriving at high altitude, with supplementary oxygen), intervention 3 (after having spent a night at high altitude)
  The impact of age and sex on medical performance during all points of testing (baseline, interventions 1-3) will be analysed by including the interactions of two variables (age and sex) with the fixed effect (representing the four time points) in the linear mixed-effect regression model described under the primary outcome. The statistical significance of the interaction will be assessed with a likelihood ratio test.
  Patient care is measured through a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT).
The correlations between psychomotor test results (PVT, BART, DSST, self-assessment of cognitive function) and medical performance during low altitude, acute and subacute high altitude exposure, measured as a composite of STAT, CALM, and TEAM scores | Baseline, intervention 1 (30 minutes after arriving at high altitude), intervention 2 (4 hours after arriving at high altitude, with supplementary oxygen), intervention 3 (after having spent a night at high altitude)
  Cognitive functions, such as measured by the psychomotor tests the investigators imply, can be impaired by high altitude exposure. The Psychomotor Vigilance Test (PVT) measures reaction speed in milliseconds. The Balloon Analogue Risk Task (BART) measures risk-taking behaviour in three numerical outcome variables. The Digit Symbol Substitution Test (DSST) measures cognitive performance and has a number of correct answers the participant found as its outcome. Participants will also self-assess their cognitive function on a scale of 1 to 10.
  The investigators will look for statistical correlations between the results of psychomotor testing (PVT, BART, DSST) and the self-assessment of cognitive capacity, and the quality of patient care at all four time points (baseline, interventions 1-3). Patient care is measured through a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT).
The correlations between vital parameters (blood pressure, heart rate, peripheral blood oxygen saturation) and medical performance during low altitude, acute and subacute high altitude exposure, measured as a composite of STAT, CALM, and TEAM scores | Baseline, intervention 1 (30 minutes after arriving at high altitude), intervention 2 (4 hours after arriving at high altitude, with supplementary oxygen), intervention 3 (after having spent a night at high altitude)
  The investigators will measure basic vital parameters of participants (blood pressure, heart rate, and peripheral blood oxygen saturation) by non-invasive means at all time points of testing (baseline, interventions 1-3). They will look for correlations between those parameters and the medical performance. Patient care is measured through a composite score comprising three previously validated scores (25% CALM, 25% TEAM, 50% STAT).

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Knapp, PD, MD, Principal Investigator — University Hospital of Bern (Inselspital), Department of Anaesthesiology and Pain Medicine
Locations (2):
- Switzerland (2):
  - Berner Simulations- und CPR-Zentrum BeSiC, Bern
  - High Altitude Research Station Jungfraujoch, Bern

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared in the primary publication(s). IPD can be made available at a reasonable request.

REFERENCES:
- [Background] Luks AM, Beidleman BA, Freer L, Grissom CK, Keyes LE, McIntosh SE, Rodway GW, Schoene RB, Zafren K, Hackett PH. Wilderness Medical Society Clinical Practice Guidelines for the Prevention, Diagnosis, and Treatment of Acute Altitude Illness: 2024 Update. Wilderness Environ Med. 2024 Mar;35(1_suppl):2S-19S. doi: 10.1016/j.wem.2023.05.013. Epub 2023 Dec 27. PMID 37833187
- [Background] McMorris T, Hale BJ, Barwood M, Costello J, Corbett J. Effect of acute hypoxia on cognition: A systematic review and meta-regression analysis. Neurosci Biobehav Rev. 2017 Mar;74(Pt A):225-232. doi: 10.1016/j.neubiorev.2017.01.019. Epub 2017 Jan 19. PMID 28111267
- [Background] Shaw DM, Cabre G, Gant N. Hypoxic Hypoxia and Brain Function in Military Aviation: Basic Physiology and Applied Perspectives. Front Physiol. 2021 May 17;12:665821. doi: 10.3389/fphys.2021.665821. eCollection 2021. PMID 34093227
- [Background] Bouak F, Vartanian O, Hofer K, Cheung B. Acute Mild Hypoxic Hypoxia Effects on Cognitive and Simulated Aircraft Pilot Performance. Aerosp Med Hum Perform. 2018 Jun 1;89(6):526-535. doi: 10.3357/AMHP.5022.2018. PMID 29789086
- [Background] Falla M, Hufner K, Falk M, Weiss EM, Vogele A, Jan van Veelen M, Weber B, Brandner J, Palma M, Dejaco A, Brugger H, Strapazzon G. Simulated Acute Hypobaric Hypoxia Effects on Cognition in Helicopter Emergency Medical Service Personnel - A Randomized, Controlled, Single-Blind, Crossover Trial. Hum Factors. 2024 Feb;66(2):404-423. doi: 10.1177/00187208221086407. Epub 2022 May 31. PMID 35640630
- [Background] Walsh JJ, Drouin PJ, King TJ, D'Urzo KA, Tschakovsky ME, Cheung SS, Day TA. Acute aerobic exercise impairs aspects of cognitive function at high altitude. Physiol Behav. 2020 Sep 1;223:112979. doi: 10.1016/j.physbeh.2020.112979. Epub 2020 May 29. PMID 32479806
- [Background] Bolmont B, Thullier F, Abraini JH. Relationships between mood states and performances in reaction time, psychomotor ability, and mental efficiency during a 31-day gradual decompression in a hypobaric chamber from sea level to 8848 m equivalent altitude. Physiol Behav. 2000 Dec;71(5):469-76. doi: 10.1016/s0031-9384(00)00362-0. PMID 11239664
- [Background] Kryskow MA, Beidleman BA, Fulco CS, Muza SR. Performance during simple and complex military psychomotor tasks at various altitudes. Aviat Space Environ Med. 2013 Nov;84(11):1147-52. doi: 10.3357/asem.3245.2013. PMID 24279227
- [Background] Narahara H, Kimura M, Suto T, Saito H, Tobe M, Aso C, Nishihara F, Saito S. Effects of cardiopulmonary resuscitation at high altitudes on the physical condition of untrained and unacclimatized rescuers. Wilderness Environ Med. 2012 Jun;23(2):161-4. doi: 10.1016/j.wem.2012.02.001. PMID 22656663
- [Background] Niederer M, Tscherny K, Burger J, Wandl B, Fuhrmann V, Kienbacher CL, Schreiber W, Herkner H, Roth D, Egger A. Influence of high altitude after a prior ascent on physical exhaustion during cardiopulmonary resuscitation: a randomised crossover alpine field experiment. Scand J Trauma Resusc Emerg Med. 2023 Oct 24;31(1):59. doi: 10.1186/s13049-023-01132-7. PMID 37875893
- [Background] Sato T, Takazawa T, Inoue M, Tada Y, Suto T, Tobe M, Saito S. Cardiorespiratory dynamics of rescuers during cardiopulmonary resuscitation in a hypoxic environment. Am J Emerg Med. 2018 Sep;36(9):1561-1564. doi: 10.1016/j.ajem.2018.01.029. Epub 2018 Jan 8. PMID 29352676
- [Background] Suto T, Saito S, Tobe M, Kanamoto M, Matsui Y. Reduction of Arterial Oxygen Saturation Among Rescuers During Cardiopulmonary Resuscitation in a Hypobaric Hypoxic Environment. Wilderness Environ Med. 2020 Mar;31(1):97-100. doi: 10.1016/j.wem.2019.10.008. Epub 2020 Feb 7. PMID 32044210
- [Background] Egger A, Niederer M, Tscherny K, Burger J, Fuhrmann V, Kienbacher C, Roth D, Schreiber W, Herkner H. Influence of physical strain at high altitude on the quality of cardiopulmonary resuscitation. Scand J Trauma Resusc Emerg Med. 2020 Mar 6;28(1):19. doi: 10.1186/s13049-020-0717-0. PMID 32143653
- [Background] Vogele A, van Veelen MJ, Dal Cappello T, Falla M, Nicoletto G, Dejaco A, Palma M, Hufner K, Brugger H, Strapazzon G. Effect of Acute Exposure to Altitude on the Quality of Chest Compression-Only Cardiopulmonary Resuscitation in Helicopter Emergency Medical Services Personnel: A Randomized, Controlled, Single-Blind Crossover Trial. J Am Heart Assoc. 2021 Dec 7;10(23):e021090. doi: 10.1161/JAHA.121.021090. Epub 2021 Dec 2. PMID 34854317
- [Background] Carballo-Fazanes A, Barcala-Furelos R, Eiroa-Bermudez J, Fernandez-Mendez M, Abelairas-Gomez C, Martinez-Isasi S, Murciano M, Fernandez-Mendez F, Rodriguez-Nunez A. Physiological demands of quality cardiopulmonary resuscitation performed at simulated 3250 meters high. Am J Emerg Med. 2020 Dec;38(12):2580-2585. doi: 10.1016/j.ajem.2019.12.048. Epub 2019 Dec 24. PMID 31911060
- [Background] Sareban M, Schiefer LM, Macholz F, Schafer L, Zangl Q, Inama F, Reich B, Mayr B, Schmidt P, Hartl A, Bartsch P, Niebauer J, Treff G, Berger MM. Endurance Athletes Are at Increased Risk for Early Acute Mountain Sickness at 3450 m. Med Sci Sports Exerc. 2020 May;52(5):1109-1115. doi: 10.1249/MSS.0000000000002232. PMID 31876668
- [Background] Mairer K, Wille M, Burtscher M. The prevalence of and risk factors for acute mountain sickness in the Eastern and Western Alps. High Alt Med Biol. 2010 Winter;11(4):343-8. doi: 10.1089/ham.2010.1039. PMID 21190503
- [Background] Berger MM, Kohne H, Hotz L, Hammer M, Schommer K, Bartsch P, Mairbaurl H. Remote ischemic preconditioning delays the onset of acute mountain sickness in normobaric hypoxia. Physiol Rep. 2015 Mar;3(3):e12325. doi: 10.14814/phy2.12325. PMID 25742960
- [Background] Roach RC, Hackett PH, Oelz O, Bartsch P, Luks AM, MacInnis MJ, Baillie JK; Lake Louise AMS Score Consensus Committee. The 2018 Lake Louise Acute Mountain Sickness Score. High Alt Med Biol. 2018 Mar;19(1):4-6. doi: 10.1089/ham.2017.0164. Epub 2018 Mar 13. PMID 29583031
- [Background] Luks AM, Swenson ER, Bartsch P. Acute high-altitude sickness. Eur Respir Rev. 2017 Jan 31;26(143):160096. doi: 10.1183/16000617.0096-2016. Print 2017 Jan. PMID 28143879
- [Background] Kammerer T, Faihs V, Hulde N, Bayer A, Hubner M, Brettner F, Karlen W, Kropfl JM, Rehm M, Spengler C, Schafer ST. Changes of hemodynamic and cerebral oxygenation after exercise in normobaric and hypobaric hypoxia: associations with acute mountain sickness. Ann Occup Environ Med. 2018 Nov 19;30:66. doi: 10.1186/s40557-018-0276-2. eCollection 2018. PMID 30479778
- [Background] Phillips L, Basnyat B, Chang Y, Swenson ER, Harris NS. Findings of Cognitive Impairment at High Altitude: Relationships to Acetazolamide Use and Acute Mountain Sickness. High Alt Med Biol. 2017 Jun;18(2):121-127. doi: 10.1089/ham.2016.0001. Epub 2017 May 16. PMID 28509579
- [Background] Issa AN, Herman NM, Wentz RJ, Taylor BJ, Summerfield DC, Johnson BD. Association of Cognitive Performance with Time at Altitude, Sleep Quality, and Acute Mountain Sickness Symptoms. Wilderness Environ Med. 2016 Sep;27(3):371-8. doi: 10.1016/j.wem.2016.04.008. Epub 2016 Jul 22. PMID 27460198
- [Background] Pun M, Guadagni V, Bettauer KM, Drogos LL, Aitken J, Hartmann SE, Furian M, Muralt L, Lichtblau M, Bader PR, Rawling JM, Protzner AB, Ulrich S, Bloch KE, Giesbrecht B, Poulin MJ. Effects on Cognitive Functioning of Acute, Subacute and Repeated Exposures to High Altitude. Front Physiol. 2018 Aug 21;9:1131. doi: 10.3389/fphys.2018.01131. eCollection 2018. PMID 30246787
- [Background] Moraga FA, Lopez I, Morales A, Soza D, Noack J. The Effect of Oxygen Enrichment on Cardiorespiratory and Neuropsychological Responses in Workers With Chronic Intermittent Exposure to High Altitude (ALMA, 5,050 m). Front Physiol. 2018 Mar 23;9:187. doi: 10.3389/fphys.2018.00187. eCollection 2018. PMID 29628892
- [Background] Meier A, Yang J, Liu J, Beitler JR, Tu XM, Owens RL, Sundararajan RL, Malhotra A, Sell RE. Female Physician Leadership During Cardiopulmonary Resuscitation Is Associated With Improved Patient Outcomes. Crit Care Med. 2019 Jan;47(1):e8-e13. doi: 10.1097/CCM.0000000000003464. PMID 30303843
- [Background] Rosenman ED, Misisco A, Olenick J, Brolliar SM, Chipman AK, Vrablik MC, Chao GT, Kozlowski SWJ, Grand JA, Fernandez R. Does team leader gender matter? A Bayesian reconciliation of leadership and patient care during trauma resuscitations. J Am Coll Emerg Physicians Open. 2021 Jan 4;2(1):e12348. doi: 10.1002/emp2.12348. eCollection 2021 Feb. PMID 33532754
- [Background] Berger MM, Husing A, Niessen N, Schiefer LM, Schneider M, Bartsch P, Jockel KH. Prevalence and knowledge about acute mountain sickness in the Western Alps. PLoS One. 2023 Sep 14;18(9):e0291060. doi: 10.1371/journal.pone.0291060. eCollection 2023. PMID 37708123
- [Background] Reid J, Stone K, Brown J, Caglar D, Kobayashi A, Lewis-Newby M, Partridge R, Seidel K, Quan L. The Simulation Team Assessment Tool (STAT): development, reliability and validation. Resuscitation. 2012 Jul;83(7):879-86. doi: 10.1016/j.resuscitation.2011.12.012. Epub 2011 Dec 23. PMID 22198422
- [Background] Nadkarni LD, Roskind CG, Auerbach MA, Calhoun AW, Adler MD, Kessler DO. The Development and Validation of a Concise Instrument for Formative Assessment of Team Leader Performance During Simulated Pediatric Resuscitations. Simul Healthc. 2018 Apr;13(2):77-82. doi: 10.1097/SIH.0000000000000267. PMID 29117092
- [Background] Florez AR, Shepard LN, Frey ME, Justice LB, Constand SE, Gilbert GE, Kessler DO, Kerrey BT, Calhoun AW. The Concise Assessment of Leader Management Tool: Evaluation of Healthcare Provider Leadership During Real-Life Pediatric Emergencies. Simul Healthc. 2023 Feb 1;18(1):24-31. doi: 10.1097/SIH.0000000000000669. Epub 2022 May 5. PMID 35533136
- [Background] Cooper S, Cant R, Porter J, Sellick K, Somers G, Kinsman L, Nestel D. Rating medical emergency teamwork performance: development of the Team Emergency Assessment Measure (TEAM). Resuscitation. 2010 Apr;81(4):446-52. doi: 10.1016/j.resuscitation.2009.11.027. Epub 2010 Feb 1. PMID 20117874
- [Background] Gawronski O, Thekkan KR, Genna C, Egman S, Sansone V, Erba I, Vittori A, Varano C, Dall'Oglio I, Tiozzo E, Chiusolo F. Instruments to evaluate non-technical skills during high fidelity simulation: A systematic review. Front Med (Lausanne). 2022 Nov 3;9:986296. doi: 10.3389/fmed.2022.986296. eCollection 2022. PMID 36405618
- [Background] Bartsch P, Swenson ER. Acute high-altitude illnesses. N Engl J Med. 2013 Oct 24;369(17):1666-7. doi: 10.1056/NEJMc1309747. No abstract available. PMID 24152275
- [Background] Stream JO, Grissom CK. Update on high-altitude pulmonary edema: pathogenesis, prevention, and treatment. Wilderness Environ Med. 2008 Winter;19(4):293-303. doi: 10.1580/07-WEME-REV-173.1. PMID 19099331
- [Background] Bartsch P, Mairbaurl H, Maggiorini M, Swenson ER. Physiological aspects of high-altitude pulmonary edema. J Appl Physiol (1985). 2005 Mar;98(3):1101-10. doi: 10.1152/japplphysiol.01167.2004. PMID 15703168